CLINICAL TRIAL: NCT03366779
Title: A Post Marketing Surveillance Study To Monitor The Early Safety And Performance Of The BARRICAID® Anular Closure Device In The Treatment Of Radicular Pain Caused By Primary Lumbar Disc Herniation
Brief Title: A Post Marketing Surveillance Study
Acronym: 6MM
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Intrinsic Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EUBARD-CP-001-6MM
Record Dates: First submitted 2017-11-28; First posted 2017-12-08 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Lumbar Disc Herniation; Annular Disc Tear; Annular Tear of Lumbar Disc
Keywords: Lumbar disc herniation, reherniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: Multicenter non-randomized device trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgery with 6mm ACD (Other): ACD medical device (non-experimental). Surgical device implantation after standard lumbar discectomy.
  Interventions: Device: 6mm annular closure device

INTERVENTIONS:
Device: 6mm annular closure device — 6MM Barricaid annular closure device implantation following standard lumbar discectomy

SUMMARY:
This study is a prospective, multi-center study to monitor the early safety and performance of one iteration of the Barricaid Anular Closure Device (ACD) - 6mm anchor width, when used as an adjunct to limited discectomy.

DETAILED DESCRIPTION:
This study is planned to collect information on use of the Barricaid ACD with an anchor width of 6mm. Other iterations of the device are made with an 8mm wide anchor. The narrower anchor was designed to optimize surgeon visualization during implantation, and has undergone all appropriate rigorous testing prior to release. Safety will be evaluated to demonstrate acceptable levels of device-related and procedure-related complications. This limited market release will allow its performance to be evaluated by examining the effects on reoperation, device deficiencies, patient pain scores and disability after discectomy with ACD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years old (male or female).
* Patients with posterior or posterolateral disc herniations at one level between L1 and S1 with radiographic confirmation of neural compression using CT and/or MRI.
* At least six (6) weeks of failed, conservative treatment prior to surgery, or requires immediate surgery to prevent permanent disability.
* Minimum posterior disc height of 5mm at the index level(s).
* Lower back pain and/or sciatica with or without spinal claudication.
* Oswestry Questionnaire score of at least 40/100 at baseline.
* VAS leg pain of at least 40/100 at baseline.
* Psychosocially, mentally and physically able to fully comply with the clinical protocol and willing to adhere to follow-up schedule and requirements.

Exclusion Criteria:

* Spondylolisthesis Grade II or higher.
* Subject requires uni or bilateral facetectomy to treat leg/back pain.
* Subject has back or non-radicular leg pain of unknown etiology.
* Prior surgery at the index lumbar level.
* Subject requiring a spine DEXA (i.e., patients with SCORE of ≥ 6) with a T Score less than -2.0 at the index level. For patients with a herniation at L5/S1, the average T score of L1-L4 shall be used.
* Subject has clinically compromised vertebral bodies at the index level(s) due to any traumatic, neoplastic, metabolic, or infectious pathology.
* Subject has sustained pathologic fractures of the vertebra or multiple fractures of the vertebra or hip.
* Subject has scoliosis of greater than ten (10) degrees (both angular and rotational).
* Any metabolic disease bone disease that has not been stabilized for at least three months (e.g., Paget's disease, osteomalacia, osteogenesis imperfecta, thyroid and/or parathyroid gland disorder, etc.).
* Subject has an active infection either systemic or local.
* Subject has cauda equina syndrome or neurogenic bowel/bladder dysfunction.
* Subject has severe arterial insufficiency of the legs (Screening on physical examination= patients with diminution or absence of dorsalis pedis or posterior tibialis pulses. If diminished or absent by palpation, then an arterial ultrasound is required with vascular plethysmography. If the absolute arterial pressure is below 50mm of Hg at the calf or ankle level, then the patient is to be excluded) or other peripheral vascular disease).
* Subject has significant peripheral neuropathy, patient defined as a patient with Type I or Type II diabetes or similar systemic metabolic condition causing decreased sensation in a stocking-like or non-radicular and non-dermatomal distribution in the lower extremities.
* Subject has insulin-dependent diabetes mellitus.
* Subject is morbidly obese (defined as a body mass index >40, or weighs more than 100 lbs over ideal body weight).
* Subject has been diagnosed with active hepatitis, AIDS, or HIV.
* Subject has been diagnosed with rheumatoid arthritis or other autoimmune disease.
* Subject has a known allergy to titanium, polyethylene or polyester materials.
* Subject is pregnant or interested in becoming pregnant in the next two (2) years.
* Subject has active tuberculosis or has had tuberculosis in the past three (3) years.
* Subject has a history of active malignancy: A patient with a history of any invasive malignancy (except non-melanoma skin cancer), unless he/she has been treated with curative intent and there have been no signs or symptoms of the malignancy for at least two (2) years.
* Subject is immunologically suppressed, received steroids >1 month over the past year.
* Currently taking anticoagulants, other than aspirin, unless the patient can be taken off the anticoagulant for surgery.
* Subject has a current chemical/alcohol dependency or significant psychosocial disturbance.
* Subject has a life expectancy of less than three (3) years.
* Subject is currently involved in another investigational study.
* Subject is incarcerated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Device stability | 3 months post implantation
  To be considered a success the subjects would require to have a lack of implant migration through 3 months after surgery

SECONDARY OUTCOMES:
Device condition, reoperation at index level and long term performance | Through 24Month post implantation
  Will be analyzed and compared to available clinical and commercial data on the Barricaid device
Visual Analog Scale - leg pain | Through 24Month post implantation
  Change in leg pain as measured using a Visual Analog Scale (VAS), on a scale of 0-100, with lower values representing better outcome.
Visual Analog scale - back pain | Through 24Month post implantation
  Change in back pain as measured using a Visual Analog Scale (VAS), on a scale of 0-100, with lower values representing better outcome.
Oswestry Disability Index | Through 24Month post implantation
  Change in function as measured using the Oswestry Disability Index (ODI)

CONTACTS AND LOCATIONS:
Locations (2):
- OLVZ Aalst, Aalst, Belgium
- Klinikum Itzehoe, Itzehoe, Germany